CLINICAL TRIAL: NCT00495859
Title: Randomized Controlled Double Blind Multi-Center Clinical Trial to Assess the Effects of Preoperative Long-Term Immunonutrition in Patients Listed for Liver Transplantation
Brief Title: Effects of Preoperative Long-Term Immunonutrition in Patients Listed for Liver Transplantation
Acronym: PROUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Prof. Peter Schemmer, MD, Dept. of surgery, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PROUD
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Newly Registered Patients for Primary Liver Transplantation
Keywords: Immunonutrition; immune enhancing diets; arginine; ω-3 fatty acids; nucleotides; liver transplantation; clinical trial
MeSH Terms: interventions — Immunonutrition Diet; Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Study group will receive formula enriched with arginine, ω-3 fatty acids, and nucleotides once daily
  Interventions: Dietary Supplement: Immunonutrition
- 2 (Active Comparator): controls receive an isocaloric isonitrogenous non-specific nutritional support
  Interventions: Dietary Supplement: food for special medical purposes (FSMP)

INTERVENTIONS:
Dietary Supplement: Immunonutrition — food for special medical purpose (FSMP)
  Other Names: ORAL IMPACT®
  Arms: 1
Dietary Supplement: food for special medical purposes (FSMP) — an isocaloric isonitrogenous non-specific nutritional support
  Other Names: IMPACT-Control Supplement
  Arms: 2

SUMMARY:
Patients with endstage liver disease characteristically are malnourished which is associated with poor outcome. Formulas enriched with arginine,ω3 fatty acids, and nucleotides potentially improve their nutritional status. This randomized placebo-controlled double blind multicenter clinical trial with longterm preoperative supplementation with such an enriched formula will evaluate evaluate effects of such formulas on patients' quality of life, survival, and posttransplant morbidities.

DETAILED DESCRIPTION:
Background. Patients with end stage liver disease characteristically are malnourished which is associated with poor outcome. Formulas enriched with arginine, ω-3 fatty acids, and nucleotides, "immunonutrients", potentially improve their nutritional status. This study is designed to evaluate the clinical outcome of long-term "immunonutrition" of patients with end-stage liver disease while on the waiting list for liver transplantation.

Methods / design. A randomized controlled double blind multi-center clinical trial with two parallel groups comprising a total of 142 newly registered patients for primary liver transplantation has been designed to assess the safety and efficacy of the long-term administration of ORAL IMPACT®, an "immunonutrient" formula, while waiting for a graft. Patients will be enrolled the day of registration on the waiting list for liver transplantation. Study ends on the day of transplantation. Primary endpoints include patients' nutritional and physiological status, as measured by mid-arm muscle area, triceps skin fold thickness, grip strength, and fatigue score, as well as patients' health related quality of life. Furthermore, patients will be followed for 12 postoperative weeks to evaluate anabolic recovery after transplantation as shown by reduced post-transplant mechanical ventilation, hospital stay, wound healing, infectious morbidities (pneumonia, intra-abdominal abscess, sepsis, line sepsis, wound infection, and urinary tract infection), acute and chronic rejection, and mortality.

Discussion. Formulas enriched with arginine, ω-3 fatty acids, and nucleotides have been proven to be beneficial in reducing postoperative infectious complications and length of hospital stay among the patients undergoing elective gastrointestinal surgery. Possible mechanisms include downregulation of the inflammatory responses to surgery and immune modulation rather than a sole nutritional effect.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 68 years of age
* Scheduled for first liver transplantation
* Written informed consent
* Protein-calorie malnutrition: Mid-arm muscle area (MAMA) <85% standard

Exclusion Criteria:

* Patients < 18 and > 68 years
* Pregnant or nursing women
* History of hypersensitivity to arginine, ω-3 fatty acids, or nucleotides
* Inability to take oral nutrition
* Patients with fulminant or subacute hepatic failure requiring urgent transplantation
* Mental condition rendering the subject incapable to understand the nature, scope, and consequences of the trial
* Simultaneous participation in another clinical trial

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
improved patients' nutritional and physiological status, fatigue score, as well as patients' health related quality of life. | while in the waiting list for liver transplantation

SECONDARY OUTCOMES:
enhanced anabolic recovery after transplantation as shown by reduced post-transplant morbidities and mortalities | the first 12 posttransplant weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schemmer, MD, Principal Investigator — Department of Surgery, Ruprecht-Karls University of Heidelberg, Germany
Locations (1):
- Department of Surgery, Ruprecht-Karls University, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Nickkholgh A, Schneider H, Encke J, Buchler MW, Schmidt J, Schemmer P. PROUD: effects of preoperative long-term immunonutrition in patients listed for liver transplantation. Trials. 2007 Aug 27;8:20. doi: 10.1186/1745-6215-8-20. PMID 17723147
- See also: Heidelberg University Hospital — http://www.klinikum.uni-heidelberg.de/
- See also: Learn more about the Department of Surgery at Ruprecht-Karls University of Heidelberg — http://www.chirurgieinfo.com